CLINICAL TRIAL: NCT03193190
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatment Combinations in Patients With Metastatic Pancreatic Ductal Adenocarcinoma (Morpheus-Pancreatic Cancer)
Brief Title: A Study of Multiple Immunotherapy-Based Treatment Combinations in Participants With Metastatic Pancreatic Ductal Adenocarcinoma (Morpheus-Pancreatic Cancer)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO39608; 2016-004126-42 (EudraCT Number)
Record Dates: First submitted 2017-06-09; First posted 2017-06-20 (Actual); Results first posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Oxaliplatin; Leucovorin; Fluorouracil; atezolizumab; cobimetinib; PEGPH20; 4-fluorobenzoyl-TN-14003; selicrelumab; Bevacizumab; Tiragolumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Cohort 1: Control (Nab-Paclitaxel and Gemcitabine) (Active Comparator): Cohort 1: Participants will receive Nab-Paclitaxel 125 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; and Gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle.
  Participants in the Cohort 1 control arm who experience disease progression will be given the option of enrolling into Cohort 2 (if open for enrollment), provided they meet eligibility criteria.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine
- Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab (Experimental): Cohort 1: Participants will receive Atezolizumab 840 mg IV infusion on Days 1 and 15 of each 28 day cycle; Nab-paclitaxel 125 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; Gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; and Selicrelumab 16 mg subcutaneous injection on Day 1 of Cycles 1-4 and every third cycle thereafter (i.e. Cycles 7, 10, 13 etc.) of each 28-day cycle.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Atezolizumab; Drug: Selicrelumab
- Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab (Experimental): Cohort 1: Participants will receive Atezolizumab 840 mg IV infusion on Days 1 and 15 of each 28 day cycle; Bevacizumab 10 mg/kg IV infusion on Days 1 and 15 of each 28 day cycle; Nab-paclitaxel 125 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; Gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Atezolizumab; Drug: Bevacizumab
- Cohort 1: Atezolizumab + Chemotherapy + AB928 (Experimental): Cohort 1: Participant will receive AB928 150 mg orally once daily on Days 1 to 28 of each 28 day cycle; Atezolizumab 840 mg IV infusion on Days 1 and 15 of each 28 day cycle; Nab-paclitaxel 125 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; Gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Atezolizumab; Drug: AB928
- Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab (Experimental): Cohort 1: Participants will receive Atezolizumab 840 mg IV infusion on Days 1 and 15 of each 28 day cycle; Tiragolumab 420 mg IV infusion on Days 1 and 15 of each 28 day cycle; Nab-paclitaxel 125 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; Gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Atezolizumab; Drug: Tiragolumab
- Cohort 2: Atezolizumab + Cobimetinib (Experimental): Cohort 2: Participants will receive Cobimetinib 60 milligrams (mg) once daily orally on Days 1-21 of each 28-day cycle; and Atezolizumab 840 mg IV infusion on Days 1 and 15 of each 28-day cycle.
  Participants who progressed on treatment may have the option of receiving Atezolizumab + RO6874281 treatment, provided they meet the eligibility criteria and the arm is open for enrollment.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- Cohort 2: Atezolizumab + PEGPH20 (Experimental): Cohort 2: Participants will receive PEGPH20 3 micrograms per kilogram (mcg/kg) IV infusion on Days 1, 8 and 15 of each 21-day cycle; and Atezolizumab 1200 mg IV infusion on Day 1 of each 21-day cycle.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Cobimetinib or Atezolizumab + RO6874281 treatment, provided they meet the eligibility criteria and the arms are open for enrollment.
  Interventions: Drug: Atezolizumab; Drug: PEGPH20
- Cohort 2: Atezolizumab + BL-8040 (Experimental): Cohort 2: Participants will receive BL-8040 1.25 milligrams per kilogram (mg/kg) subcutaneously (SC) on Days 1-5 of the first week, followed by combination treatment consisting of BL-8040 1.25 mg/kg SC three times a week on non-consecutive days and Atezolizumab 1200 mg IV infusion on Day 1 of each 21-day cycle.
  Participants who progressed on treatment may have the option of receiving Atezolizumab + Cobimetinib or Atezolizumab + RO6874281 treatment, provided they meet the eligibility criteria and the arms are open for enrollment.
  Interventions: Drug: Atezolizumab; Drug: BL-8040
- Cohort 2: Atezolizumab + RO6874281 every 2 weeks (Experimental): Cohort 2: Participants will receive Atezolizumab 840 mg IV infusion on days 1 and 15 of each 28 day cycle; RO6874281 will be administered 10 mg by IV infusion on day 1 and 15 mg on days 8, 15, and 22 for cycle 1 (28 day cycle). RO6874281 will be administered 15 mg by IV infusion on days 1 and 15 of each subsequent 28 day cycle.
  Participants who progressed on treatment may have the option of receiving Atezolizumab + Cobimetinib, provided they meet the eligibility criteria and the arm is open for enrollment.
  Interventions: Drug: Atezolizumab; Drug: RO6874281
- Cohort 2: Atezolizumab + RO6874281 every 3 weeks (Experimental): Cohort 2: Participants will receive Atezolizumab 1200 mg IV infusion on Day 1 of each 21 day cycle; and RO6874281 10 mg by IV infusion on day 1 of each 21 day cycle.
  Participants who progressed on treatment may have the option of receiving Atezolizumab + Cobimetinib, provided they meet the eligibility criteria and the arm is open for enrollment.
  Interventions: Drug: Atezolizumab; Drug: RO6874281
- Cohort 2: Control (Nab-Paclitaxel and Gemcitabine or mFOLFOX6) (Active Comparator): Cohort 2: Participants who progressed on a prior fluoropyrimidine-based regimen will receive Nab-paclitaxel 125 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; and Gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle.
  Participants who progressed on a prior gemcitabine-based regimen will receive 5-fluorouracil, leucovorin, and oxaliplatin (mFOLFOX6). Participants will receive Oxaliplatin 85 mg/m^2 IV on Days 1 and 15 of each 28 day cycle; Leucovorin 400 mg/m^2 IV on Days 1 and 15 of each 28 day cycle; Fluorouracil 400 mg/m^2 IV push on Days 1 and 15 of each 28 day cycle; and Fluorouracil 2400 mg/m^2 IV continuous infusion over 46 hours on Days 1 and 2 and on Days 15 and 16 of each 28 day cycle.
  Participants who progressed on treatment, may have the option of receiving Atezolizumab + Cobimetinib or Atezolizumab + RO6874281 treatment, provided they meet the eligibility criteria and the arms are open for enrollment.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil
- Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab (Experimental): Cohort 1: Participants will receive Tocilizumab 8 mg/kg IV infusion on Day 1 of each 28 day cycle; Atezolizumab 1680 mg IV infusion on Day 1 of each 28 day cycle; Nab-paclitaxel 125 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle; and Gemcitabine 1000 mg/m^2 IV infusion on Days 1, 8, and 15 of each 28 day cycle.
  Interventions: Drug: Nab-Paclitaxel; Drug: Gemcitabine; Drug: Atezolizumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: Nab-Paclitaxel — Nab-Paclitaxel will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + AB928; Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Cohort 1: Control (Nab-Paclitaxel and Gemcitabine); Cohort 2: Control (Nab-Paclitaxel and Gemcitabine or mFOLFOX6)
Drug: Gemcitabine — Gemcitabine will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + AB928; Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Cohort 1: Control (Nab-Paclitaxel and Gemcitabine); Cohort 2: Control (Nab-Paclitaxel and Gemcitabine or mFOLFOX6)
Drug: Oxaliplatin — Oxaliplatin will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 2: Control (Nab-Paclitaxel and Gemcitabine or mFOLFOX6)
Drug: Leucovorin — Leucovorin will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 2: Control (Nab-Paclitaxel and Gemcitabine or mFOLFOX6)
Drug: Fluorouracil — Fluorouracil will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 2: Control (Nab-Paclitaxel and Gemcitabine or mFOLFOX6)
Drug: Atezolizumab — Atezolizumab will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + AB928; Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Cohort 2: Atezolizumab + BL-8040; Cohort 2: Atezolizumab + Cobimetinib; Cohort 2: Atezolizumab + PEGPH20; Cohort 2: Atezolizumab + RO6874281 every 2 weeks; Cohort 2: Atezolizumab + RO6874281 every 3 weeks
Drug: Cobimetinib — Cobimetinib will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 2: Atezolizumab + Cobimetinib
Drug: PEGPH20 — PEGPH20 will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 2: Atezolizumab + PEGPH20
Drug: BL-8040 — BL-8040 will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 2: Atezolizumab + BL-8040
Drug: Selicrelumab — Selicrelumab will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab
Drug: Bevacizumab — Bevacizumab will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab
Drug: RO6874281 — RO6874281 will be administered as per the schedule specified in the respective arm
  Arms: Cohort 2: Atezolizumab + RO6874281 every 2 weeks; Cohort 2: Atezolizumab + RO6874281 every 3 weeks
Drug: AB928 — AB928 will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + AB928
Drug: Tiragolumab — Tiragolumab will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab
Drug: Tocilizumab — Tocilizumab will be administered as per the schedule specified in the respective arm.
  Arms: Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab

SUMMARY:
A Phase Ib/II, open-label, multicenter, randomized study designed to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of immunotherapy-based treatment combinations in participants with metastatic Pancreatic Ductal Adenocarcinoma (PDAC).

Two cohorts will be enrolled in parallel in this study: Cohort 1 will consist of patients who have received no prior systemic therapy for metastatic PDAC, and Cohort 2 will consist of patients who have received one line of prior systemic therapy for PDAC. In each cohort, eligible patients will be assigned to one of several treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically or cytologically confirmed metastatic pancreatic ductal adenocarcinoma
* For patients in Cohort 1: no prior systemic treatment for PDAC
* For patients in Cohort 2: disease progression during administration of either 5-FU- or gemcitabine-based first-line chemotherapy
* Life expectancy greater than or equal to 3 months
* Availability of a representative tumor specimen that is suitable for determination of programmed death-ligand 1 (PD-L1) and/or additional biomarker status via central testing
* Measurable disease (at least one target lesion) according to RECIST v1.1
* Adequate hematologic and end-organ function test results
* Tumor accessible for biopsy
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs, as outlined for each specific treatment arm
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as outlined for each specific treatment arm

Exclusion Criteria:

* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring drainage procedure (i.e., more than one time per month)
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Positive human immunodeficiency (HIV) test at screening or at any time prior to screening
* Active hepatitis B or C virus infection or active tuberculosis
* Severe infection within 4 weeks prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplantation
* History of malignancy other than pancreatic carcinoma within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (12):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Helen Diller Fam Comp Can Ctr, San Francisco, California
  - Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut
  - Lombardi Cancer Center, Georgetown University, Washington D.C., District of Columbia
  - Uni of Chicago Medical Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - MorristownMedicalCenter, Morristown, New Jersey
  - Columbia University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Universitätsklinikum Essen, Essen, Germany
- Japan (3):
  - National Cancer Center Hospital East, Chiba
  - Kanagawa Cancer Center, Kanagawa
  - National Cancer Center Hospital, Tokyo
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hosp. G. U Gregorio Marañón, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid

REFERENCES:
- [Derived] Ko AH, Kim KP, Siveke JT, Lopez CD, Lacy J, O'Reilly EM, Macarulla T, Manji GA, Lee J, Ajani J, Alsina Maqueda M, Rha SY, Lau J, Al-Sakaff N, Allen S, Lu D, Shemesh CS, Gan X, Cha E, Oh DY. Atezolizumab Plus PEGPH20 Versus Chemotherapy in Advanced Pancreatic Ductal Adenocarcinoma and Gastric Cancer: MORPHEUS Phase Ib/II Umbrella Randomized Study Platform. Oncologist. 2023 Jun 2;28(6):553-e472. doi: 10.1093/oncolo/oyad022. PMID 36940261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 341 participants with metastatic pancreatic ductal adenocarcinoma (PDAC) took part in the study from 05 Jul 2017 to 27 Feb 2025. The study included participants in 2 cohorts: Cohort 1: received no prior systemic therapy for metastatic PDAC & Cohort 2: received 1 prior line of systemic therapy for PDAC. Multiple combination therapies were compared against common control(s) in Cohorts 1 and 2.
Pre-assignment Details: Eligible participants from both cohorts were assigned to one of several treatment arms in Stage 1. Cohort 2 participants with disease progression (PD), loss of clinical benefit, or unacceptable toxicity in Stage 1 were eligible for a different treatment combination in Stage 2. The study is considered "Completed" because all the pre-planned study activities and analyses have been performed.
Groups:
- Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine): Participants received nab-paclitaxel, 125 milligrams/meter square (mg/m^2), intravenous (IV) infusion and gemcitabine ,1000 mg/m^2, IV infusion on Days 1, 8, and 15 of each cycle until unacceptable toxicity or PD (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab: Participants received atezolizumab, 840 mg, IV infusion on Days 1 and 15 of each cycle along with nab-paclitaxel, 125 mg/m^2 and gemcitabine, 1000 mg/m^2, also administered as IV infusion on Days 1, 8, and 15 of each cycle. Participants also received selicrelumab, 16 mg, subcutaneous (SC) injection on Day 1 of Cycles 1-4 and every third cycle thereafter (i.e. Cycles 7, 10, 13 etc.) of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab: Participants received atezolizumab, 840 mg, and bevacizumab, 10 milligrams/kilograms (mg/kg), IV infusion on Days 1 and 15 of each cycle along with nab-paclitaxel 125 mg/m^2, and gemcitabine, 1000 mg/m^2 also administered as IV infusion on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928: Participants received AB928, 150 mg, orally, once daily (QD) on Days 1 to 28 of each cycle; atezolizumab 840 mg, IV infusion on Days 1 and 15 of each cycle and nab-paclitaxel, 125 mg/m^2, and gemcitabine, 1000 mg/m^2, also administered as IV infusion, on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab: Participants received atezolizumab, 840 mg and tiragolumab, 420 mg, IV infusion on Days 1 and 15 of each cycle along with nab-paclitaxel, 125 mg/m^2 and gemcitabine, 1000 mg/m^2, also administered as IV infusion on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab: Participants received atezolizumab, 1680 mg and tocilizumab, 8 mg/kg, IV infusion on Days 1 of each cycle along with nab-paclitaxel, 125 mg/m^2 and gemcitabine, 1000 mg/m^2, also administered as IV infusion on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]): Participants who progressed on a prior gemcitabine-based regimen received mFOLFOX6 which is oxaliplatin, 85 mg/m^2 and leucovorin, 400 mg/m^2 as IV infusion, and 5-fluorouracil, 400 mg/m^2, IV push on Days 1 and 15 of each cycle along with 5-fluorouracil, 2400 mg/m^2, IV continuous infusion on Days 1, 2, 15 and 16 of each cycle until unacceptable toxicity or PD (1 cycle=28 days).
- Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine): Participants who progressed on a prior fluoropyrimidine-based regimen received nab-paclitaxel, 125 mg/m^2 and gemcitabine, 1000 mg/m^2, also administered as IV infusion on Days 1, 8, and 15 of each cycle until unacceptable toxicity or PD (1 cycle=28 days).
- Stage 1 Cohort 2: Atezolizumab + BL-8040: Participants received BL-8040, 1.25 mg/kg, SC injection on Days 1-5 of the first week, as priming treatment, and thereafter three times a week (Days 1, 3, 5, 8, 10, 12, 15, 17, and 19) along with atezolizumab, 1200 mg, IV infusion on Day 1 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 1 Cohort 2: Atezolizumab + Cobimetinib: Participants received atezolizumab, 840 mg, IV infusion on Days 1 and 15 of each cycle and cobimetinib 60 mg, orally, QD on Days 1-21 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 2: Atezolizumab + PEGPH20: Participants received atezolizumab, 1200 mg, IV infusion on Day 1 of each cycle and PEGPH20, 3 micrograms per kilogram (µg/kg), IV infusion on Days 1, 8 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 1 Cohort 2: Atezolizumab + RO6874281 Every 3 Weeks (Q3W): Participants received atezolizumab, 1200 mg, IV infusion and RO6874281, 10 mg, IV infusion on Day 1 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 1 Cohort 2: Atezolizumab + RO6874281 Every 2 Weeks (Q2W): Participants received atezolizumab, 840 mg, IV infusion on Days 1 and 15 of each cycle and RO6874281, 10 mg, IV infusion on Day 1 and 15 mg on Days 8, 15, and 22 of Cycle 1 and thereafter 15 mg on Days 1 and 15 of subsequent cycles until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 2 Cohort 2: Atezolizumab + Cobimetinib: Participants in Cohort 2 control and experimental arms (other than atezolizumab + cobimetinib) who experienced PD, loss of clinical benefit, or unacceptable toxicity during Stage 1 and met the eligibility criteria to enroll in Stage 2 received atezolizumab, 840 mg, IV infusion on Days 1 and 15 of each cycle and cobimetinib, 60 mg, orally, QD on Days 1-21 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 2 Cohort 2: Atezolizumab + RO6874281 Q3W: Participants in cohort 2 control and experimental arms (other than atezolizumab + RO6874281 Q3W) who experienced PD, loss of clinical benefit, or unacceptable toxicity during Stage 1 received atezolizumab, 1200 mg, IV infusion and RO6874281, 10 mg, as IV infusion on Day 1 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 2 Cohort 2: Atezolizumab + RO6874281 Q2W: Participants in cohort 2 control and experimental arms (other than atezolizumab + RO6874281 Q2W) who experienced PD, loss of clinical benefit, or unacceptable toxicity during Stage 1 received atezolizumab, 840 mg, IV infusion on Days 1 and 15 of each cycle and RO6874281, 10 mg, IV infusion on Day 1 and 15 mg on Days 8, 15, and 22 of Cycle 1 and thereafter 15 mg on Days 1 and 15 of subsequent cycles until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
Period: Stage 1
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Every 3 Weeks (Q3W) | Stage 1 Cohort 2: Atezolizumab + RO6874281 Every 2 Weeks (Q2W) | Stage 2 Cohort 2: Atezolizumab + Cobimetinib | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q2W
Started | 35 | 9 | 25 | 16 | 42 | 31 | 25 | 25 | 16 | 15 | 71 | 16 | 15 | 0 | 0 | 0
Safety Population (Safety population included all participants who received any amount of study treatment.) | 32 | 9 | 25 | 15 | 41 | 30 | 23 | 23 | 15 | 14 | 66 | 15 | 14 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 35 | 9 | 25 | 16 | 42 | 31 | 25 | 25 | 16 | 15 | 71 | 16 | 15 | 0 | 0 | 0
Not completed — Arm Terminated by Sponsor | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 22 | 8 | 23 | 14 | 34 | 28 | 19 | 21 | 14 | 10 | 59 | 14 | 14 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not Specified | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 3 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 1 | 0 | 2 | 0 | 3 | 2 | 2 | 4 | 9 | 1 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Every 3 Weeks (Q3W) | Stage 1 Cohort 2: Atezolizumab + RO6874281 Every 2 Weeks (Q2W) | Stage 2 Cohort 2: Atezolizumab + Cobimetinib | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q2W
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 6 | 1
Safety Population (Safety population included all participants who received any amount of study treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 6 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 15 | 6 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 4 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population included all randomized participants.
Groups:
- Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine): Participants received nab-paclitaxel, 125 mg/m^2, IV infusion and gemcitabine, 1000 mg/m^2, IV infusion on Days 1, 8, and 15 of each cycle until unacceptable toxicity or PD (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab: Participants received atezolizumab, 840 mg, IV infusion on Days 1 and 15 of each cycle along with nab-paclitaxel, 125 mg/m^2 and gemcitabine, 1000 mg/m^2, also administered as IV infusion on Days 1, 8, and 15 of each cycle. Participants also received selicrelumab, 16 mg, SC injection on Day 1 of Cycles 1-4 and every third cycle thereafter (i.e. Cycles 7, 10, 13 etc.) of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab: Participants received atezolizumab, 840 mg, and bevacizumab, 10 mg/kg, IV infusion on Days 1 and 15 of each cycle along with nab-paclitaxel 125 mg/m^2, and gemcitabine, 1000 mg/m^2 also administered as IV infusion on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928: Participants received AB928, 150 mg, orally, QD on Days 1 to 28 of each cycle; atezolizumab 840 mg, IV infusion on Days 1 and 15 of each cycle and nab-paclitaxel, 125 mg/m^2, and gemcitabine, 1000 mg/m^2, also administered as IV infusion, on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1 Cohort 2: Atezolizumab + PEGPH20: Participants received atezolizumab, 1200 mg, IV infusion on Day 1 of each cycle and PEGPH20, 3 µg/kg, IV infusion on Days 1, 8 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W: Participants received atezolizumab, 1200 mg, IV infusion and RO6874281, 10 mg, IV infusion on Day 1 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W: Participants received atezolizumab, 840 mg, IV infusion on Days 1 and 15 of each cycle and RO6874281, 10 mg, IV infusion on Day 1 and 15 mg on Days 8, 15, and 22 of Cycle 1 and thereafter 15 mg on Days 1 and 15 of subsequent cycles until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Total: Total of all reporting groups
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W | Total
Number analyzed (Participants) | 35 | 9 | 25 | 16 | 42 | 31 | 25 | 25 | 16 | 15 | 71 | 16 | 15 | 341
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 15 | 6 | 13 | 11 | 26 | 11 | 9 | 20 | 8 | 9 | 49 | 8 | 8 | 193
  65-84 years | 20 | 3 | 12 | 5 | 16 | 20 | 16 | 5 | 8 | 6 | 22 | 8 | 7 | 148
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 7 | 8 | 12 | 11 | 14 | 11 | 5 | 5 | 28 | 9 | 7 | 134
  Male | 22 | 5 | 18 | 8 | 30 | 20 | 11 | 14 | 11 | 10 | 43 | 7 | 8 | 207
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 12
  Not Hispanic or Latino | 33 | 9 | 23 | 16 | 36 | 30 | 25 | 24 | 16 | 15 | 68 | 16 | 14 | 325
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Asian | 12 | 1 | 5 | 8 | 8 | 12 | 11 | 6 | 8 | 4 | 21 | 6 | 3 | 105
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 9
  White | 18 | 4 | 16 | 7 | 30 | 15 | 14 | 19 | 7 | 9 | 43 | 10 | 11 | 203
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 5 | 1 | 2 | 0 | 3 | 3 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 20

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percentage of Participants With Objective Response (OR), as Determined by Investigator According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: OR was defined as a complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart during Stage 1 as determined by the investigator using RECIST v.1.1. Objective response rate (ORR) was defined as the percentage of participants with OR. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of target lesions, taking as reference the baseline SOD. 95% confidence intervals (CI) for rates were constructed using Clopper-Pearson method. Percentages have been rounded off.
Time Frame: Up to 33.3 months
Population: Efficacy population included participants in the safety population who received at least one dose of study drug and who had at least one baseline and one on-study tumor assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W
Number analyzed (Participants) | 32 | 9 | 25 | 15 | 41 | 30 | 23 | 23 | 14 | 14 | 66 | 15 | 14
percentage of participants | 37.5 [21.10 to 56.31] | 55.6 [21.20 to 86.30] | 48.0 [27.80 to 68.69] | 26.7 [7.79 to 55.10] | 31.7 [18.08 to 48.09] | 30.0 [14.73 to 49.40] | 8.7 [1.07 to 28.04] | 0 [0.00 to 14.82] | 0 [0.00 to 23.16] | 0 [0.00 to 23.16] | 6.1 [1.68 to 14.80] | 0 [0.00 to 21.80] | 7.1 [0.18 to 33.87]
Statistical Analysis 1: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Test type: Superiority; Difference in ORR = 18.06, 95% CI 2-sided [-25.60 to 61.71]
Statistical Analysis 2: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Test type: Superiority; Difference in ORR = 10.50, 95% CI 2-sided [-18.85 to 39.85]
Statistical Analysis 3: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928; Test type: Superiority; Difference in ORR = -10.83, 95% CI 2-sided [-43.70 to 22.03]
Statistical Analysis 4: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Test type: Superiority; Difference in Overall Response Rates = -5.79, 95% CI 2-sided [-30.58 to 18.99]
Statistical Analysis 5: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Test type: Superiority; Difference in ORR = -7.50, 95% CI 2-sided [-34.19 to 19.19]
Statistical Analysis 6: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + BL-8040; Test type: Superiority; Difference in ORR = -8.70, 95% CI 2-sided [-25.96 to 8.57]
Statistical Analysis 7: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + Cobimetinib; Test type: Superiority; Difference in Overall Response Rates = -8.70, 95% CI 2-sided [-25.96 to 8.57]
Statistical Analysis 8: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + PEGPH20; Test type: Superiority; Difference in ORR = -2.64, 95% CI 2-sided [-18.44 to 13.17]
Statistical Analysis 9: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W; Test type: Superiority; Difference in ORR = -8.70, 95% CI 2-sided [-25.72 to 8.33]
Statistical Analysis 10: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W; Test type: Superiority; Difference in ORR = -1.55, 95% CI 2-sided [-25.04 to 21.93]

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including abnormal laboratory values or abnormal clinical test results), symptoms, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product.
Time Frame: Up to 33.3 months
Population: Safety population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W | Stage 2 Cohort 2: Atezolizumab + Cobimetinib | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q2W
Number analyzed (Participants) | 32 | 9 | 25 | 15 | 41 | 30 | 23 | 23 | 15 | 14 | 66 | 15 | 14 | 14 | 6 | 1
Participants | 32 | 9 | 24 | 15 | 41 | 30 | 22 | 23 | 15 | 14 | 65 | 15 | 14 | 14 | 6 | 0

3. Secondary Outcome: Stage 1: Progression-Free Survival (PFS), as Determined by Investigator According to RECIST v1.1
Description: PFS was defined as the time from study treatment initiation to the first occurrence of documented PD, as determined by the investigator according to RECIST v1.1 or death from any cause, whichever occurs first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Kaplan-Meier (K-M) method was used to estimate PFS.
Time Frame: Up to 33.3 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W
Number analyzed (Participants) | 32 | 9 | 25 | 15 | 41 | 30 | 23 | 23 | 14 | 14 | 66 | 15 | 14
months | 6.11 [5.13 to 9.92] | 4.04 [3.02 to 6.97] | 7.18 [5.03 to 9.82] | 8.21 [5.91 to 11.10] | 5.82 [4.40 to 7.52] | 5.39 [4.17 to 8.21] | 2.76 [1.45 to 5.52] | 2.53 [1.77 to 4.04] | 1.64 [1.41 to 1.87] | 1.28 [1.15 to 1.84] | 1.51 [1.38 to 2.56] | 1.38 [1.38 to 2.66] | 1.46 [1.31 to 1.58]
Statistical Analysis 1: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Test type: Superiority; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.48 to 2.64]
Statistical Analysis 2: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Test type: Superiority; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.66 to 2.08]
Statistical Analysis 3: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928; Test type: Superiority; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.29 to 1.23]
Statistical Analysis 4: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.67 to 1.89]
Statistical Analysis 5: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Test type: Superiority; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.61 to 1.87]
Statistical Analysis 6: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + BL-8040; Test type: Superiority; Hazard Ratio (HR) = 2.13, 95% CI 2-sided [0.96 to 4.75]
Statistical Analysis 7: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + Cobimetinib; Test type: Superiority; Hazard Ratio (HR) = 3.63, 95% CI 2-sided [1.54 to 8.57]
Statistical Analysis 8: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + PEGPH20; Test type: Superiority; Hazard Ratio (HR) = 1.15, 95% CI 2-sided [0.68 to 1.92]
Statistical Analysis 9: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W; Test type: Superiority; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [0.72 to 3.05]
Statistical Analysis 10: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W; Test type: Superiority; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [0.84 to 3.06]

4. Secondary Outcome: Stage 1: Overall Survival (OS), as Determined by Investigator According to RECIST v1.1
Description: OS was defined as the time from randomization to death from any cause. K-M method was used to estimate OS.
Time Frame: Up to 33.3 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W
Number analyzed (Participants) | 32 | 9 | 25 | 15 | 41 | 30 | 23 | 23 | 14 | 14 | 66 | 15 | 14
months | 14.55 [9.99 to 16.16] | 9.03 [3.42 to 16.13] | 13.34 [9.10 to 15.21] | 16.49 [9.59 to 19.71] | 13.34 [9.43 to 21.59] | 11.20 [8.21 to 17.94] | 6.77 [6.34 to 9.66] | 8.31 [4.11 to 13.04] | 4.47 [3.12 to 7.06] | 4.24 [1.84 to 6.97] | 7.06 [4.07 to 8.38] | 4.70 [3.81 to 11.04] | 7.33 [4.86 to 11.60]
Statistical Analysis 1: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Test type: Superiority; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.59 to 3.00]
Statistical Analysis 2: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Test type: Superiority; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.71 to 2.29]
Statistical Analysis 3: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928; Test type: Superiority; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.45 to 1.74]
Statistical Analysis 4: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.58 to 1.68]
Statistical Analysis 5: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.59 to 1.84]
Statistical Analysis 6: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + BL-8040; Test type: Superiority; Hazard Ratio (HR) = 2.04, 95% CI 2-sided [0.87 to 4.77]
Statistical Analysis 7: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + Cobimetinib; Test type: Superiority; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [0.60 to 2.94]
Statistical Analysis 8: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + PEGPH20; Test type: Superiority; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.48 to 1.60]
Statistical Analysis 9: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W; Test type: Superiority; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.68 to 3.36]
Statistical Analysis 10: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W; Test type: Superiority; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.44 to 2.02]

5. Secondary Outcome: Stage 1: OS Rate at Month 6
Description: OS was defined as the time from randomization to death from any cause. OS rate at 6 months was defined as the percentage of participants who did not experience death from any cause at 6 months from randomization. K-M method was used to estimate OS. Percentages have been rounded off.
Time Frame: Month 6
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W
Number analyzed (Participants) | 32 | 9 | 25 | 15 | 41 | 30 | 23 | 23 | 14 | 14 | 66 | 15 | 14
percentage of participants | 87.07 [75.23 to 98.91] | 55.56 [23.09 to 88.02] | 83.48 [68.67 to 98.28] | 80.00 [59.76 to 100.00] | 72.55 [58.72 to 86.37] | 86.67 [74.50 to 98.83] | 78.76 [60.06 to 97.46] | 53.45 [30.72 to 76.19] | 27.78 [1.17 to 54.39] | 41.96 [14.01 to 69.91] | 51.97 [39.29 to 64.65] | 43.33 [17.35 to 69.32] | 50.00 [23.81 to 76.19]
Statistical Analysis 1: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Test type: Superiority; Difference in Event Free Rate = -31.51, 95% CI 2-sided [-66.07 to 3.04]
Statistical Analysis 2: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Test type: Superiority; Difference in Event Free Rate = -3.59, 95% CI 2-sided [-22.55 to 15.37]
Statistical Analysis 3: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928; Test type: Superiority; Difference in Event Free Rate = -7.07, 95% CI 2-sided [-30.52 to 16.38]
Statistical Analysis 4: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Test type: Superiority; Difference in Event Free Rate = -14.52, 95% CI 2-sided [-32.72 to 3.68]
Statistical Analysis 5: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Test type: Superiority; Difference in Event Free Rate = -0.40, 95% CI 2-sided [-17.38 to 16.57]
Statistical Analysis 6: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + BL-8040; Test type: Superiority; Difference in Event Free Rate = -50.98, 95% CI 2-sided [-83.51 to -18.46]
Statistical Analysis 7: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + Cobimetinib; Test type: Superiority; Difference in Event Free Rate = -36.80, 95% CI 2-sided [-70.43 to -3.18]
Statistical Analysis 8: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + PEGPH20; Test type: Superiority; Difference in Event Free Rate = -26.79, 95% CI 2-sided [-49.39 to -4.20]
Statistical Analysis 9: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W; Test type: Superiority; Difference in Event Free Rate = -35.43, 95% CI 2-sided [-67.44 to -3.42]
Statistical Analysis 10: Comparison: Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) vs Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W; Test type: Superiority; Difference in Event Free Rate = -28.76, 95% CI 2-sided [-60.94 to 3.42]

6. Secondary Outcome: Stage 1: Duration of Response (DOR), as Determined by Investigator According to RECIST v1.1
Description: DOR was defined as time from first occurrence of a documented OR until the time of documented PD or death from any cause, whichever occurs first as determined by investigator assessment using RECIST v1.1. DOR was calculated for participants who had a best confirmed OR of CR/PR. CR=the disappearance of all target lesions or any pathological lymph nodes (whether target or non-target) having a reduction in short axis to <10 mm. PR=at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. PD=at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum on the study including baseline (nadir). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. K-M method was used to estimate DOR.
Time Frame: Up to 33.3 months
Population: Efficacy population included participants in the safety population who received at least one dose of study drug and who had at least one baseline and one on-study tumor assessment. Overall number analyzed included participants with OR i.e responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W
Number analyzed (Participants) | 12 | 5 | 12 | 4 | 13 | 9 | 2 | 0 | 0 | 0 | 4 | 0 | 1
months | 5.40 [3.94 to 8.21] | 3.35 [2.56 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. | 8.18 [6.34 to 8.74] | 4.85 [2.86 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. | 4.47 [3.58 to 10.12] | 5.65 [4.53 to 10.84] | 3.37 [2.83 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. |  |  |  | 8.15 [5.32 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. |  | 6.14 [NA to NA] — The 95% CI was not estimable due to an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab; Test type: Superiority; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.24 to 3.51]
Statistical Analysis 2: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab; Test type: Superiority; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.23 to 1.60]
Statistical Analysis 3: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928; Test type: Superiority; Hazard Ratio (HR) = 1.56, 95% CI 2-sided [0.44 to 5.47]
Statistical Analysis 4: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.35 to 2.44]
Statistical Analysis 5: Comparison: Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) vs Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab; Test type: Superiority; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.24 to 1.93]

7. Secondary Outcome: Stage 1: Percentage of Participants With Disease Control (DC), as Determined by Investigator According to RECIST v1.1
Description: DC was defined as stable disease (SD) for ≥ 12 weeks or a CR or PR, as determined by the investigator according to RECIST v1.1 Disease control rate (DCR) was defined as the percentage of participants with DC. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) have a reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the SOD of target lesions, taking as reference the baseline SOD. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Percentages have been rounded off.
Time Frame: Up to 33.3 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W
Number analyzed (Participants) | 32 | 9 | 25 | 15 | 41 | 30 | 23 | 23 | 14 | 14 | 66 | 15 | 14
percentage of participants | 81.3 [63.56 to 92.79] | 55.6 [21.20 to 86.30] | 64.0 [42.52 to 82.03] | 66.7 [38.38 to 88.18] | 61.0 [44.50 to 75.80] | 66.7 [47.19 to 82.71] | 30.4 [13.21 to 52.92] | 34.8 [16.38 to 57.27] | 0 [0.00 to 23.16] | 0 [0.00 to 23.16] | 18.2 [9.76 to 29.61] | 0 [0.00 to 21.80] | 7.1 [0.18 to 33.87]

ADVERSE EVENTS:
Time Frame: Up to 33.3 months
Description: Safety population included all participants who received any amount of study treatment.
Arm/Group | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) | Stage 1 Cohort 2: Atezolizumab + BL-8040 | Stage 1 Cohort 2: Atezolizumab + Cobimetinib | Stage 1 Cohort 2: Atezolizumab + PEGPH20 | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W | Stage 2 Cohort 2: Atezolizumab + Cobimetinib | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q3W | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q2W
All-Cause Mortality (participants affected / at risk) | 23/32 | 8/9 | 23/25 | 14/15 | 34/41 | 28/30 | 19/23 | 21/23 | 14/15 | 11/14 | 60/66 | 14/15 | 14/14 | 14/14 | 5/6 | 1/1
Serious Adverse Events (participants affected / at risk) | 13/32 | 8/9 | 17/25 | 4/15 | 19/41 | 12/30 | 10/23 | 12/23 | 4/15 | 8/14 | 30/66 | 7/15 | 2/14 | 7/14 | 2/6 | 0/1
Other Adverse Events (participants affected / at risk) | 32/32 | 9/9 | 23/25 | 15/15 | 40/41 | 30/30 | 21/23 | 23/23 | 15/15 | 13/14 | 65/66 | 15/15 | 14/14 | 13/14 | 6/6 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) (N=32) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab (N=9) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab (N=25) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 (N=15) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab (N=41) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab (N=30) | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) (N=23) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) (N=23) | Stage 1 Cohort 2: Atezolizumab + BL-8040 (N=15) | Stage 1 Cohort 2: Atezolizumab + Cobimetinib (N=14) | Stage 1 Cohort 2: Atezolizumab + PEGPH20 (N=66) | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W (N=15) | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W (N=14) | Stage 2 Cohort 2: Atezolizumab + Cobimetinib (N=14) | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q3W (N=6) | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q2W (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic duct obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sweat gland infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolic cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle cerebral artery stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudocellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angiodysplasia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Cohort 1 : Control (Chemotherapy: Nab-Paclitaxel and Gemcitabine) (N=32) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Selicrelumab (N=9) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Bevacizumab (N=25) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + AB928 (N=15) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tiragolumab (N=41) | Stage 1 Cohort 1: Atezolizumab + Chemotherapy + Tocilizumab (N=30) | Stage 1 Cohort 2: Control (5-fluorouracil + Leucovorin + Oxaliplatin [mFOLFOX6]) (N=23) | Stage 1 Cohort 2: Control (Nab-Paclitaxel and Gemcitabine) (N=23) | Stage 1 Cohort 2: Atezolizumab + BL-8040 (N=15) | Stage 1 Cohort 2: Atezolizumab + Cobimetinib (N=14) | Stage 1 Cohort 2: Atezolizumab + PEGPH20 (N=66) | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q3W (N=15) | Stage 1 Cohort 2: Atezolizumab + RO6874281 Q2W (N=14) | Stage 2 Cohort 2: Atezolizumab + Cobimetinib (N=14) | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q3W (N=6) | Stage 2 Cohort 2: Atezolizumab + RO6874281 Q2W (N=1)
Anaemia (Blood and lymphatic system disorders) | 14 (15) | 4 (5) | 10 (11) | 9 (9) | 13 (19) | 6 (6) | 4 (4) | 6 (7) | 3 (3) | 2 (2) | 8 (9) | 1 (1) | 1 (1) | 3 (3) | 2 (3) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 10 (13) | 1 (1) | 4 (8) | 1 (5) | 7 (13) | 9 (12) | 6 (6) | 4 (5) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 5 (5) | 2 (2) | 8 (12) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central serous chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Halo vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (5) | 0 (0) | 3 (3) | 2 (2) | 7 (8) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (10) | 3 (3) | 5 (5) | 2 (2) | 11 (12) | 4 (5) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 9 (10) | 3 (3) | 1 (1) | 3 (4) | 1 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (6) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 12 (12) | 2 (2) | 5 (5) | 4 (4) | 10 (11) | 10 (10) | 7 (7) | 5 (5) | 5 (6) | 2 (2) | 10 (13) | 6 (7) | 7 (8) | 1 (4) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (16) | 2 (2) | 9 (14) | 4 (6) | 15 (18) | 11 (13) | 2 (2) | 4 (4) | 2 (2) | 5 (9) | 11 (12) | 4 (4) | 3 (3) | 6 (9) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (20) | 7 (7) | 9 (12) | 7 (9) | 21 (23) | 16 (19) | 10 (12) | 9 (12) | 5 (5) | 7 (8) | 20 (23) | 6 (7) | 9 (12) | 2 (6) | 3 (4) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 2 (2) | 5 (5) | 3 (3) | 3 (4) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (9) | 3 (6) | 10 (15) | 2 (2) | 8 (10) | 6 (10) | 7 (10) | 4 (4) | 2 (2) | 5 (8) | 11 (14) | 4 (4) | 4 (6) | 4 (5) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (7) | 0 (0) | 3 (4) | 5 (5) | 6 (10) | 3 (5) | 6 (6) | 4 (4) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 10 (14) | 6 (7) | 1 (2) | 2 (2) | 0 (0)
Face oedema (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 18 (22) | 5 (7) | 11 (16) | 3 (4) | 23 (25) | 7 (7) | 5 (5) | 9 (9) | 10 (11) | 5 (6) | 21 (22) | 5 (5) | 6 (8) | 2 (2) | 2 (2) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 5 (7) | 2 (2) | 2 (2) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (21) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 11 (17) | 4 (4) | 7 (7) | 4 (4) | 16 (19) | 9 (10) | 2 (3) | 7 (9) | 1 (1) | 2 (2) | 22 (26) | 2 (2) | 2 (2) | 5 (5) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 11 (13) | 5 (6) | 3 (4) | 3 (3) | 14 (19) | 2 (2) | 1 (1) | 5 (11) | 2 (2) | 5 (5) | 7 (9) | 7 (12) | 10 (12) | 2 (3) | 3 (4) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular icterus (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 2 (7) | 0 (0) | 0 (0) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (25) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 8 (8) | 3 (4) | 6 (8) | 6 (7) | 7 (7) | 14 (15) | 0 (0) | 6 (6) | 2 (2) | 3 (3) | 7 (7) | 5 (8) | 5 (7) | 0 (0) | 1 (2) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 4 (4) | 5 (6) | 6 (7) | 7 (7) | 11 (14) | 1 (1) | 7 (8) | 1 (1) | 7 (7) | 8 (9) | 6 (10) | 6 (8) | 0 (0) | 1 (2) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 2 (2) | 2 (2) | 4 (5) | 5 (5) | 2 (2) | 1 (2) | 7 (7) | 2 (2) | 3 (3) | 8 (8) | 4 (5) | 5 (5) | 3 (3) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (2) | 1 (2) | 0 (0) | 3 (5) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (9) | 4 (5) | 8 (11) | 5 (6) | 10 (16) | 18 (22) | 3 (3) | 8 (9) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 3 (4) | 4 (7) | 4 (6) | 11 (17) | 16 (20) | 2 (3) | 4 (5) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 5 (5) | 2 (2) | 6 (6) | 1 (1) | 7 (7) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 4 (4) | 2 (3) | 3 (3) | 4 (5) | 4 (9) | 10 (11) | 0 (0) | 5 (7) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 13 (14) | 3 (4) | 10 (14) | 7 (7) | 14 (15) | 9 (10) | 9 (10) | 3 (3) | 4 (4) | 3 (3) | 14 (15) | 4 (4) | 3 (3) | 4 (5) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 5 (5) | 2 (2) | 3 (4) | 5 (5) | 0 (0) | 3 (3) | 4 (6) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 4 (4) | 2 (2) | 3 (3) | 3 (5) | 3 (4) | 2 (2) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 1 (1) | 3 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 7 (8) | 2 (2) | 3 (3) | 2 (2) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (5) | 6 (6) | 1 (1) | 5 (6) | 4 (6) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 16 (18) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 6 (7) | 5 (6) | 0 (0) | 5 (6) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (11) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 3 (3) | 0 (0) | 5 (7) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 45 (50) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 6 (7) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 4 (4) | 2 (3) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2) | 4 (7) | 3 (3) | 4 (5) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 0 (0) | 5 (7) | 1 (2) | 4 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 8 (8) | 0 (0) | 10 (11) | 0 (0) | 11 (11) | 4 (4) | 2 (3) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 3 (4) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (9) | 2 (2) | 3 (3) | 4 (4) | 5 (5) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 2 (3) | 3 (3) | 0 (0) | 6 (6) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Testicular disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 3 (3) | 6 (9) | 1 (1) | 8 (9) | 4 (5) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 6 (10) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 6 (6) | 1 (1) | 12 (12) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 8 (8) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 6 (6) | 2 (2) | 6 (8) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14) | 3 (3) | 4 (4) | 4 (4) | 14 (14) | 9 (9) | 1 (1) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 5 (7) | 5 (6) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (8) | 1 (1) | 5 (8) | 6 (7) | 15 (22) | 9 (11) | 0 (0) | 5 (5) | 3 (8) | 1 (1) | 3 (3) | 2 (2) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 1 (1) | 7 (7) | 5 (5) | 10 (11) | 4 (4) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 3 (5) | 8 (8) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolism venous (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1) | 9 (13) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 5 (6) | 2 (2) | 0 (0) | 1 (3) | 1 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT03193190/Prot_SAP_000.pdf